CLINICAL TRIAL: NCT01639911
Title: STM-01: Phase I EffTox Study of Aurora A Kinase Inhibitor Alisertib (MLN8237) Given in Combination With Selective VEGFR Inhibitor Pazopanib (Votrient) for Therapy of Solid Tumors
Brief Title: Phase I Study of MLN8237 and Pazopanib in Patients With Solid Tumors
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: University of Illinois at Chicago (Other)
Collaborators: Millennium Pharmaceuticals, Inc. (Industry)
Responsible Party: Principal Investigator, Arkadiusz Dudek, MD, Professor, University of Illinois at Chicago
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2013-0100; X14011 (Other: Millennium); 2013-0100 (Other: University of Illinois at Chicago (UIC) Office for the Protection of Research Subjects (OPRS))
Record Dates: First submitted 2012-03-26; First posted 2012-07-13 (Estimated); Last update posted 2019-07-22 (Actual); Status verified 2019-07

CONDITIONS: Malignant Neoplasm of Breast; CNS Malignancy; Malignant Neoplasm of Gastrointestinal Tract; Genitourinary Neoplasms Malignancy and Gender Unspecified; Head and Neck Neoplasms; Melanoma; Malignant Neoplasm of Thorax
Keywords: malignant solid tumor; advanced non-hematologic
MeSH Terms: conditions — Breast Neoplasms; Central Nervous System Neoplasms; Gastrointestinal Neoplasms; Head and Neck Neoplasms; Melanoma | interventions — MLN 8237; pazopanib

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes

ARMS (1):
- Treated Patients with Solid Tumor (Experimental): Patients will receive alisertib orally twice a day for the first 7 days of a 21 day cycle. Patients will also receive pazopanib orally once a day continuously. Treatment continues until disease progression, unacceptable toxicity or patient refusal. The study consists of two components which are the dose finding component and optimally tolerated dose extension with pharmacokinetics component.
  Interventions: Drug: Alisertib; Drug: Pazopanib

INTERVENTIONS:
Drug: Alisertib — Alisertib at the assigned dose by mouth (PO) twice a day for 7 days beginning on day 1 of a 21 day cycle.
  Other Names: MLN8237
Drug: Pazopanib — Pazopanib at the assigned dose once a day continuously for the duration of treatment.
  Other Names: Votrient

SUMMARY:
This phase I trial using the EffTox design will evaluate activity and safety of alisertib, an Aurora A kinase inhibitor, when given in combination with the selective VEGFR inhibitor pazopanib in patients with advanced, previously treated non-hematologic solid tumors.

ELIGIBILITY:
Inclusion Criteria:

1. Diagnosis of advanced non-hematologic solid tumor malignancy, including, but not limited to breast, lung, colon, pancreatic, head and neck, kidney or sarcoma that has failed or become intolerant to standard therapy and is no longer likely to respond to such therapy. Note: The MTD for pazopanib monotherapy in patients with hepatocellular cancer was found to be 600 mg daily therefore enrollment for these patients will be limited to pazopanib dose levels at or below 600 mg.
2. Measurable disease per RECIST version 1.1
3. Age ≥ 18 years
4. ECOG PS of 0-2
5. Prior systemic chemotherapy, immunotherapy, or biological therapy is allowed; however prior use of study drugs in combination is not allowed.

   Time since prior therapy and the first dose of study drug
   * At least 21 days since previous antineoplastic therapy
   * At least 42 days since previous nitrosoureas or mitomycin-C
   * At least 42 days since exposure to fully human monoclonal antibodies
   * At least 28 days since previous chimeric monoclonal antibodies
   * At least 14 days since noncytotoxic small molecule drugs (eg tyrosine kinase inhibitors such as Tarceva® and hormonal agents such as Femara®)
   * At least 21 days since previous radiation therapy
   * At least 14 days since prior major surgery (defined as a surgery involving a risk to the life of the patient; specifically: an operation upon an organ within the cranium, chest, abdomen, or pelvic cavity)
   * At least 3 months since prior autologous transplant
6. Must have recovered from the reversible effects (≤ grade 1 CTCAE) of previous anti-cancer treatment prior to study registration
7. Adequate organ function within 14 days of study registration defined as:

   * Absolute neutrophil count (ANC) > 1500/mm^3
   * Hemoglobin > 9 g/dL (Values must be obtained without need for myeloid growth factor or platelet transfusion support within 14 days, however, erythrocyte growth factor is allowed as per published ASCO guidelines)
   * Platelets > 100,000/mm^3 (Values must be obtained without need for myeloid growth factor or platelet transfusion support within 14 days, however, erythrocyte growth factor is allowed as per published ASCO guidelines)
   * Total bilirubin Within normal limits
   * SGOT (AST) and SGPT (ALT) ≤1.5 X ULN
   * If liver metastases present: Total bilirubin Within normal limits and SGOT (AST) and SGPT (ALT) ≤ 3.0 X ULN
   * Glomerular filtration rate (GFR) ≥ 40 mL/minute
   * Urine dipstick for proteinuria < 1+ within 1 week prior to registration (If urine dipstick ≥ 1, then a 24-hour urine protein must demonstrate ≤ 1 gram protein in 24 hours to participate in study)

   NOTE: Patients with liver metastases will be allowed to participate with SGOT (AST) and SGPT (ALT) of up to 3.0 times the upper limits of normal.
8. Patient must be able to take oral medication and to maintain a fast as required for 2 hrs before and 2 hrs after alisertib administration
9. Female patient is either post-menopausal or surgically sterilized or willing to use an acceptable method of birth control (ie, a hormonal contraceptive, intra-uterine device, diaphragm with spermicide, condom with spermicide, or abstinence) for the duration of the study and for 4 months after the last dose of alisertib.
10. Male patient agrees to use an acceptable method for contraception during the entire study treatment period through 4 months after the last dose of alisertib.
11. Voluntary written consent before performance of any study-related procedure not part of normal medical care, with the understanding that consent may be withdrawn by the patient at any time without prejudice to future medical care.

Exclusion Criteria:

1. Untreated or symptomatic CNS metastases
2. Radiation therapy to more than 25% of the bone marrow. Whole pelvic radiation is is considered to be over 25%.
3. Prior allogeneic bone marrow transplantation
4. ≥ Grade 2 peripheral neuropathy within 14 days before enrollment
5. Known history of uncontrolled sleep apnea and other conditions that could result in excessive daytime sleepiness, such as severe chronic obstructive pulmonary disease; requirement for supplemental oxygen.
6. Requirement for constant admin. of proton pump inhibitor, H2 antagonist, or pancreatic enzymes. Intermittent uses of antacids or H2 antagonists are allowed as described in the protocol.
7. Systemic infection requiring IV antibiotics within 14 days preceding the 1st dose of study drug, or other severe infection.
8. Myocardial infarction within 6 months prior to enrollment or has New York Heart Association (NYHA) Class II, III or IV heart failure, uncontrolled angina, severe uncontrolled ventricular arrhythmias, or electrocardiographic evidence of acute ischemia or active conduction system abnormalities requiring therapy. Prior to study entry, any ECG abnormality at Screening has to be documented by the investigator as not medically relevant.
9. Pregnant or breast-feeding. Pazopanib is Pregnancy Category D - known teratogenic potential. Confirmation that the subject is not pregnant must be established by a negative serum beta-human chorionic gonadotropin (beta-hCG) pregnancy test result obtained during screening. Pregnancy testing is not required for post-menopausal or surgically sterilized women.
10. Patient has received other investigational drugs with 14 days before enrollment
11. Serious medical or psychiatric illness in the opinion of the researcher that would likely interfere with participation in this clinical study.
12. Other severe acute or chronic medical or psychiatric condition, including uncontrolled diabetes, malabsorption, resection of the pancreas or upper small bowel, requirement for pancreatic enzymes, any condition that would modify small bowel absorption of oral medications, or laboratory abnormality that may increase the risk associated with study participation or investigational product administration or may interfere with the interpretation of study results and, in the judgment of the investigator, would make the patient inappropriate for enrollment in this study.
13. Treatment with clinically significant enzyme inducers, such as the enzyme-inducing antiepileptic drugs phenytoin, carbamazepine or phenobarbital, or rifampin, rifabutin, rifapentine or St. John's wort within 14 days prior to the first dose of alisertib and during the study.
14. Treatment should be avoided (however not prohibited) with strong UGT inhibitors such as atazanavir, gemfibrozil, indinavir, ketoconazole, Silybum marianum (milk thistle), Valeriana officinalis (garden valerian) or inducers such as carbamazepine, nicotine, Orthosiphon stamineus within 14 days prior to the first dose of alisertib and during the study.
15. Known history of human immunodeficiency virus (HIV) infection, hepatitis B, or hepatitis C. Testing is not required in the absence of clinical findings or suspicion.
16. Recent (within 6 months) arterial thromboembolic events, including transient ischemic attack (TIA), cerebrovascular accident (CVA), unstable angina, or myocardial infarction (MI). Patients with clinically significant peripheral artery disease are ineligible.
17. History of thrombotic or hemorrhagic disorders, not receiving chronic daily treatment with aspirin (>325 mg/day) or non-steriodal anti-inflammatory agents know to inhibit platelet function. Treatment with dipyridamole (persantine), ticlopidine (Ticlid), clopidogrel (Plavix) and/or cilostazol (Pletal).
18. Use of simvastatin is not recommended but not prohibited. The concomitant use of pazopanib and simvastatin increases the risk of ALT elevations. Discontinue simvastatin if possible to decrease risk of transaminases elevation from pazopanib. There are insufficient data available to assess the risk of alternative statins. If it must be continued, monitor liver function closely and follow dosing guidelines.
19. History of abdominal fistula, gastrointestinal perforation, or intra abdominal abscess within 28 days prior to beginning study treatment
20. Clinically significant gastrointestinal abnormalities that may affect absorption of investigational product including, but not limited to:

    * Ongoing nausea or vomiting of any severity
    * > grade 1 diarrhea
    * Malabsorption syndrome
    * Major resection of stomach or small bowel
21. Inability to swallow oral medications or inability to take nothing by mouth except water and prescribed medications for 2 hours before and 2 hours after each dose of alisertib.
22. Abnormalities on 12-lead electrocardiogram (ECG) considered by the investigator to be clinical significant or baseline prolongation of the rate-corrected QT interval (e.g., repeated demonstration of QTc interval > 450 milliseconds)
23. Poorly controlled hypertension [defined as systolic blood pressure (SBP) of ≥140 mmHg or diastolic blood pressure (DBP) of ≥ 90mmHg]. Note: Initiation or adjustment of antihypertensive medication(s) is permitted prior to study entry. The mean SBP / DBP values from each blood pressure assessment must be < 140/90mmHg in order for a subject to be eligible for the study.
24. History of cerebrovascular accident, pulmonary embolism or untreated deep venous thrombosis (DVT) within the past 6 months. Note: Subjects with recent DVT who have been treated with therapeutic anti-coagulating agents for at least 6 weeks are eligible. Patients receiving Coumadin must be transition to low molecular weight heparin and treated for at least 14 days prior to the first dose of study drug.
25. Presence of any non-healing wound, fracture, or ulcer within 28 days prior to the first dose of study drug
26. Evidence of active bleeding or bleeding diathesis
27. Known endobronchial lesions or involvement of large pulmonary vessels by tumor or centrally located pulmonary cavitating lesion
28. Hemoptysis (> ½ teaspoon of bright red blood per episode) within 6 weeks of first dose of study drug
29. Unable or unwilling to discontinue use of prohibited medications list in Section 6.5 for at least 14 days prior to the first dose of study drug and for the duration of the study
30. Known immediate or delayed hypersensitivity reaction or idiosyncrasy to drugs chemically related to pazopanib or alisertib

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 28 (Actual)
Dates: Start 2013-08-14 (Actual); Primary Completion 2016-07-28 (Actual); Study Completion 2016-07-28 (Actual)

PRIMARY OUTCOMES:
Optimally Tolerated Dose | At end of Cycle 1 (approximately Day 21)
  Complete all planned treatment for cycle 1 (defined as 14 doses of alisertib and daily pazopanib) without dose limiting toxicity and are able to start cycle 2 with no more than a 2 week delay.

SECONDARY OUTCOMES:
Toxicity Profile | Within 30 days of Last Treatment Dose
  Adverse events which occur after taking at least one dose of study treatment with either alisertib and/or pazopanib.

CONTACTS AND LOCATIONS:
Overall Officials: Arkadiusz Z. Dudek, M.D., Principal Investigator — University of Illinois at Chicago
Locations (1):
- University of Illinois Cancer Center, Chicago, Illinois, United States

REFERENCES:
- [Derived] Shah HA, Fischer JH, Venepalli NK, Danciu OC, Christian S, Russell MJ, Liu LC, Zacny JP, Dudek AZ. Phase I Study of Aurora A Kinase Inhibitor Alisertib (MLN8237) in Combination With Selective VEGFR Inhibitor Pazopanib for Therapy of Advanced Solid Tumors. Am J Clin Oncol. 2019 May;42(5):413-420. doi: 10.1097/COC.0000000000000543. PMID 30973373